CLINICAL TRIAL: NCT05413590
Title: Description of Physical Activity Effect on Neuromuscular Fatigue of Older People
Acronym: ACTIFS-AGE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollments
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21CH033; ANSM (Other: 2021-A01228-33)
Record Dates: First submitted 2022-02-10; First posted 2022-06-10 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Aging; Fatigue
Keywords: cardiovascular function; neuromuscular function; V02max
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Young, Active group (Active Comparator): From 18 to 35 years old.
  The subjects will be considered as active if after completion of the Global Physical Activity Questionnaire (GPAQ), the subjects count:
  * at least 20 minutes of vigorous physical activity per day for 3 or more days per week OR
  * at least 30 minutes of moderate physical activity or walking per day for 5 or more days per week OR
  * At least 5 days of walking and moderate or vigorous physical activity, reaching a minimum of 600 Metabolic Equivalent of Task (MET)-minutes per week
  Interventions: Other: Questionnaires completion; Other: Isometric forces; Other: Energy cost
- Young, sedentary group (Active Comparator): From 18 to 35 years old. Subjects who are below these thresholds will be considered as sedentary. To avoid including a subject who recently changed his lifestyle (sedentary becoming active or vice versa), the investigator will ensure the subject kept this physical activity level (expressed using the GPAQ) constant for the last 5 years.
  Interventions: Other: Questionnaires completion; Other: Isometric forces; Other: Energy cost
- Old, Active group (Active Comparator): From 65 to 80 years old.
  The subjects will be considered as active if after completion of the Global Physical Activity Questionnaire (GPAQ), the subjects count:
  * at least 20 minutes of vigorous physical activity per day for 3 or more days per week OR
  * at least 30 minutes of moderate physical activity or walking per day for 5 or more days per week OR
  * At least 5 days of walking and moderate or vigorous physical activity, reaching a minimum of 600 MET-minutes per week
  Interventions: Other: Questionnaires completion; Other: Isometric forces; Other: Energy cost
- Old sedentary group (Active Comparator): From 65 to 80 years old. Subjects who are below these thresholds will be considered as sedentary. To avoid including a subject who recently changed his lifestyle (sedentary becoming active or vice versa), the investigator will ensure the subject kept this physical activity level (expressed using the GPAQ) constant for the last 5 years.
  Interventions: Other: Questionnaires completion; Other: Isometric forces; Other: Energy cost
- Very old, Active group (Active Comparator): From 81 years old.
  The subjects will be considered as active if after completion of the Global Physical Activity Questionnaire (GPAQ), the subjects count:
  * at least 20 minutes of vigorous physical activity per day for 3 or more days per week OR
  * at least 30 minutes of moderate physical activity or walking per day for 5 or more days per week OR
  * At least 5 days of walking and moderate or vigorous physical activity, reaching a minimum of 600 MET-minutes per week
  Interventions: Other: Questionnaires completion; Other: Isometric forces; Other: Energy cost
- Very old sedentary group (Active Comparator): From 81 years old. Subjects who are below these thresholds will be considered as sedentary. To avoid including a subject who recently changed his lifestyle (sedentary becoming active or vice versa), the investigator will ensure the subject kept this physical activity level (expressed using the GPAQ) constant for the last 5 years.
  Interventions: Other: Questionnaires completion; Other: Isometric forces; Other: Energy cost

INTERVENTIONS:
Other: Questionnaires completion — Cognitive tests, completing questionnaires, balance test, measuring cardiac variability and post-ischemic hyperemia. Assessments of neuromuscular function on a semi-recumbent ergometric bicycle.
Other: Isometric forces — Measurement of the maximum isometric forces of the knee flexors, the plantar flexors of the ankle and the grip strength of the hand.
Other: Energy cost — Measurement of feet pressure and measurement of the energy cost. Maximum test on an endocycle (classic) to determine VO2max.

SUMMARY:
There is a decrease in cardiovascular and neuromuscular functions, which leads to reduced performance with advancing age. Physical activity provides health benefits, prevents and treats cardiovascular and neuromuscular disease. The aim of this project is to describe cardiovascular and neuromuscular function in active and sedentary subjects of different ages.

DETAILED DESCRIPTION:
With advancing age, there is a decrease in cardiovascular and neuromuscular functions, which leads to reduced performance and increases the likelihood that older people will lose their independence. Physical activity provides health benefits, prevents and treats cardiovascular and neuromuscular disease. Indeed, recent data support the idea that it is fitness level, not age that explains physiological responses to exercise. However, although there are data about how quickly cardiovascular and neuromuscular functions decline throughout life, less is known on the extent physical activity can help mitigate the loss of these functions. The aim of this project is therefore to describe cardiovascular and neuromuscular function in active and sedentary subjects of different ages.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 35 for the young group, between 65 and 80 for the old group and over 80 for the very old group.
* Signed consent for the study obtained
* Subject affiliated or entitled to a social security scheme

Exclusion Criteria:

* Pathology or surgical intervention causing a locomotor disorder
* Neurological, cardiovascular or psychological pathology
* Participants will be excluded if resting or exercise ECG responses show any abnormality, or if resting Heart Rate (HR) > 100 bmp, resting blood pressure > 144 (systolic) / 95 (diastolic) mmHg, pulmonary and or cardiac disease that could affect the health of the participant (arrhythmias and stroke)
* Mini-Mental State Examination score < 20 (>80 years old)
* Significant change in the amount of physical practice over the last 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Maximal voluntary contraction (MVC) of the knee extensor muscle measurement | At 48 hours
  Maximal isometric force (maximal voluntary contraction, MVC) of the knee extensor muscle measured before and after an incremental test on a bicycle ergometer

SECONDARY OUTCOMES:
Voluntary activation measurement (%) | At 48 hours
  The level of voluntary activation will be determined by the force increment obtained following stimulation performed during a condition of the muscle in a state of maximum contraction.
Maximal voluntary contraction (MVC) of the plantar flexor muscle measurement | At 48 hours
  Maximal isometric force (maximal voluntary contraction, MVC) of the knee extensor muscle measured before and after an incremental test on a bicycle ergometer
Maximal voluntary contraction (MVC) of the hand grip measurement | At 48 hours
  Maximal isometric force (maximal voluntary contraction, MVC) of the knee extensor muscle measured before and after an incremental test on a bicycle ergometer
Cardiac variability(ms) | At 48 hours
  24-hour measurement with an ECG holter for 24 hours.
Muscle oxygenation (%) | At 48 hours
  This is measured by a NIRS20 (near infrared spectroscopy, Oxysoft, Artinis, TheNetherlands)
Balance test (s) | At 48 hours
  This test, performed in unipedal support, consists of asking the subject to hold the unipedal position for as long as possible, on the lower limb of his choice.
Test of Get-up-and-Go (s) | At 48 hours
  For test of Get-up-and-Go, participants will be asked to stand from a seated position, walk 3 meters at their usual pace, turn around, walk back to the chair, and sit down.
  Measured in seconds when performing test.
Reaction force on the ground for each step (N) | At 72 hours
  First, a maximum pace walking speed and a comfort speed will be measured in a corridor using photoelectric cells. Then, a biomechanical analysis of walking at several speeds (comfort walking, 2.5, 4 and 5.5 km/h) will be performed on an instrumented treadmill (Treadmetrix, Park City, Utah, United States). This treadmill allows the analysis of the reaction forces on the ground during the strides while controlling the speed of the walk. Each step will last approximately 30 seconds.
Maximal oxygen consumption (VO2max) during an effort test on a cycloergometer | At 72 hours
Functional Assessment of Chronic Illness Therapy (FACIT) questionnaire | At inclusion
  Score from 0 to 52
Quality of life via the SF-36 questionnaire | At inclusion
  This questionnaire is composed of 12 questions representing the eight most relevant domains to describe and evaluate quality of life. Score ranges from 0 to 100, with a higher score defining a more favorable health state.

CONTACTS AND LOCATIONS:
Overall Officials: LEONARD FEASSON, PHD, Principal Investigator — Centre Hospitalier Universitaire de Saint Etienne; Guillaume MILLET, PhD, Study Chair — UNIVERSITE DE SAINT ETIENNE
Locations (1):
- Chu de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luneau E, Rozand V, Murias JM, Millet GY. Effect of Habitual Physical Activity on Strength Loss and Fatigability in Old and Very Old Men. Scand J Med Sci Sports. 2025 Dec;35(12):e70176. doi: 10.1111/sms.70176. PMID 41343292